CLINICAL TRIAL: NCT02148068
Title: Roux-en-y Gastric Bypass Versus Sleeve Gastrectomy - Analysis of the Disparate Effects on Body Composition and Associated Comorbidity Resolution
Brief Title: Changes in Body Composition Following Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Peter Nau (Other)
Responsible Party: Sponsor-Investigator, Peter Nau, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201310819
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Obesity
Keywords: Obesity; Bariatric Surgery; Roux-en-y Gastric Bypass; Sleeve Gastrectomy
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Bariatric Surgery - Gastric Bypass: This population will undergo a laparoscopic roux-en-y gastric bypass
  Interventions: Procedure: Bariatric Surgery
- Bariatric Surgery - Sleeve Gastrectomy: This group will undergo a laparoscopic sleeve gastrectomy
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — Patients enrolled will undergo either a laparoscopic Roux-en-y Gastric Bypass or laparoscopic Sleeve Gastrectomy. The determination of which operation performed will be made independent of patients' enrollment in the study.

SUMMARY:
Obesity is an important public health issue worldwide. In the United States, the percentage of overweight and obese adults increased from 47 and 15%, respectively, to 69 and 36% in the last 40 years. Medically supervised attempts at weight loss are fraught with failures and recidivism. Surgical approaches to this important issue are both durable and effective. The gold standard approach to the surgical treatment of obesity and the attendant medical comorbidities is the laparoscopic roux-en-y gastric bypass (RYGB) and the laparoscopic sleeve gastrectomy (LSG). The mechanisms by which these two operations work and the associated side effects are not completely understood. It is established that the RYGB induces changes in both the fatty tissue mass (FTM) and lean body mass (LBM) post-operatively. This is associated with decreases in bone mineral density, basal metabolic rate, and potentially the ability to maintain weight loss. There is only incomplete information on the influence that the LSG has on body composition. This study proposes an evaluation of the changes in body composition that occurs following these two disparate operations. Using serial measurements by the BodPod and collecting information on the patients' dietary intake, exercise habits and comorbidity resolution, this study will help to better define the influence that the LSG has on body composition. It is hypothesized that the addition of a malabsorptive component will result in increased speed weight loss and overall weight loss which will have a negative impact in the preservation of lean tissue mass for the patient. This information can then be used by bariatric surgeons to better cater the surgical procedure and post-operative plan to the patient's body make up and medical comorbidities.

DETAILED DESCRIPTION:
Procedures

* All patients will undergo a bariatric surgery. The decision to undergo weight loss surgery and the operation chosen will both occur independent of and prior to enrollment in the study. The University of Iowa is a Bariatric Center of Excellence with three active, board-certified bariatric surgeons.
* Serial BodPod examinations will be performed on each patient. The BodPod is a commercially available device produced by Cosmed. It uses whole-body densitometry to determine body composition. To do this, it takes small changes in the volume of air in the BodPod chamber and records the associated changes in pressure. The pressure change typically goes unnoticed and is equivalent to the change in pressure while moving from the first floor to the second floor in an elevator. The entire process takes approximately five minutes with two minutes spent within the machine. The computer will then use mathematical formulas to calculate various body composition values.
* Laboratory analysis - There is a battery of labs that are ordered in both the pre-operative and post-operative time frame. These labs are ordered independent of the patient's participation in the study. These labs are ordered to assist in the management of the patient's medical comorbidities and to assess for adequate nutritional intake. These labs will also be recorded in the research database to assist in quantifying the degree of resolution of medical comorbidities.
* Queries on nutritional intake and exercise will be made at each post-operative appointment. The intake of protein is an important variable and may influence maintenance of lean tissue mass. Exercise is an important component of the post-bariatric weight loss program. This also will influence the changes in lean tissue mass.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will have a BMI greater than 35 kg/m2 and a medical comorbidity or 40 kg/m2
* Individuals must have voluntarily initiated a surgical consultation for weight loss surgery
* Individuals must have completed a medical supervised weight loss program

Exclusion Criteria:

* Failure to adequately complete the pre-screening and educational program necessary to proceed with bariatric surgery
* Those who are or become pregnant
* Individuals with severe claustrophobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population consists of individuals who meet the NIH consensus statement for the surgical treatment of obesity. These individuals will have a BMI greater than 35 kg/m2 and a medical comorbidity or 40 kg/m2. These subjects will have voluntarily initiated a consultation for bariatric surgery and completed the pre-bariatric surgery weight management program. After failing this program, the patients will undergo surgical consultation for bariatric surgery. It is only after this consultation that the subjects will be approached for enrollement in the study.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2014-05; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Body Composition | Pre-op, 6 months and 12 months post-op
  Using the BodPod machine produced by Cosmed, changes in lean tissue mass and fatty tissue mass following either the laparoscopic roux-en-y gastric bypass or the laparoscopic sleeve gastrectomy will be assessed.

SECONDARY OUTCOMES:
Comorbidity resolution | pre-op, 6 months post-op, 12 months post-op
  Assess for correlations between the changes in body composition and the resolution of medical comorbidities when comparing the LSG and RYGB. This will be done using changes in medication regimen and changes in physical findings and laboratory values such as blood pressure and HbA1c.
Protein intake and lean tissue mass | Pre-op, 6 months post-op, 12 months post-op
  Assess for correlation between the preservation of lean tissue mass and daily protein intake and whether the type of operation (roux-en-y gastric bypass and sleeve gastrectomy) plays a role.
Exercise and lean tissue mass preservation | Pre-op, 6 months post-op, 12 months post-op
  Test for a correlation between the changes in body composition and the amount of physical activity the patient takes part in and whether this is influenced by the type of procedure the patient had (roux-en-y gastric bypass versus sleeve gastrectomy).

CONTACTS AND LOCATIONS:
Overall Officials: Peter N Nau, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu FB. Resolved: there is sufficient scientific evidence that decreasing sugar-sweetened beverage consumption will reduce the prevalence of obesity and obesity-related diseases. Obes Rev. 2013 Aug;14(8):606-19. doi: 10.1111/obr.12040. Epub 2013 Jun 13. PMID 23763695
- [Background] Popkin BM, Adair LS, Ng SW. Global nutrition transition and the pandemic of obesity in developing countries. Nutr Rev. 2012 Jan;70(1):3-21. doi: 10.1111/j.1753-4887.2011.00456.x. PMID 22221213
- [Background] Kautiainen S, Rimpela A, Vikat A, Virtanen SM. Secular trends in overweight and obesity among Finnish adolescents in 1977-1999. Int J Obes Relat Metab Disord. 2002 Apr;26(4):544-52. doi: 10.1038/sj.ijo.0801928. PMID 12075582
- [Background] Heude B, Lafay L, Borys JM, Thibult N, Lommez A, Romon M, Ducimetiere P, Charles MA. Time trend in height, weight, and obesity prevalence in school children from Northern France, 1992-2000. Diabetes Metab. 2003 Jun;29(3):235-40. doi: 10.1016/s1262-3636(07)70032-0. PMID 12909811
- [Background] Jackson-Leach R, Lobstein T. Estimated burden of paediatric obesity and co-morbidities in Europe. Part 1. The increase in the prevalence of child obesity in Europe is itself increasing. Int J Pediatr Obes. 2006;1(1):26-32. doi: 10.1080/17477160600586614. PMID 17902212
- [Background] Schauer PR, Kashyap SR, Wolski K, Brethauer SA, Kirwan JP, Pothier CE, Thomas S, Abood B, Nissen SE, Bhatt DL. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med. 2012 Apr 26;366(17):1567-76. doi: 10.1056/NEJMoa1200225. Epub 2012 Mar 26. PMID 22449319
- [Background] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Background] Himpens J, Cadiere GB, Bazi M, Vouche M, Cadiere B, Dapri G. Long-term outcomes of laparoscopic adjustable gastric banding. Arch Surg. 2011 Jul;146(7):802-7. doi: 10.1001/archsurg.2011.45. Epub 2011 Mar 21. PMID 21422330
- [Background] Jackson TD, Hutter MM. Morbidity and effectiveness of laparoscopic sleeve gastrectomy, adjustable gastric band, and gastric bypass for morbid obesity. Adv Surg. 2012;46:255-68. doi: 10.1016/j.yasu.2012.05.002. PMID 22873044
- [Background] Moize V, Andreu A, Rodriguez L, Flores L, Ibarzabal A, Lacy A, Jimenez A, Vidal J. Protein intake and lean tissue mass retention following bariatric surgery. Clin Nutr. 2013 Aug;32(4):550-5. doi: 10.1016/j.clnu.2012.11.007. Epub 2012 Nov 14. PMID 23200926
- [Background] Chaston TB, Dixon JB, O'Brien PE. Changes in fat-free mass during significant weight loss: a systematic review. Int J Obes (Lond). 2007 May;31(5):743-50. doi: 10.1038/sj.ijo.0803483. Epub 2006 Oct 31. PMID 17075583
- [Background] Tsai S. Importance of lean body mass in the oncologic patient. Nutr Clin Pract. 2012 Oct;27(5):593-8. doi: 10.1177/0884533612457949. Epub 2012 Aug 16. PMID 22898746
- [Background] Guillet C, Masgrau A, Walrand S, Boirie Y. Impaired protein metabolism: interlinks between obesity, insulin resistance and inflammation. Obes Rev. 2012 Dec;13 Suppl 2:51-7. doi: 10.1111/j.1467-789X.2012.01037.x. PMID 23107259
- [Background] de Aquino LA, Pereira SE, de Souza Silva J, Sobrinho CJ, Ramalho A. Bariatric surgery: impact on body composition after Roux-en-Y gastric bypass. Obes Surg. 2012 Feb;22(2):195-200. doi: 10.1007/s11695-011-0500-4. PMID 21881836
- [Background] Carey DG, Pliego GJ, Raymond RL, Skau KB. Body composition and metabolic changes following bariatric surgery: effects on fat mass, lean mass and basal metabolic rate. Obes Surg. 2006 Apr;16(4):469-77. doi: 10.1381/096089206776327378. PMID 16608613